CLINICAL TRIAL: NCT05429385
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Phase I Clinical Study to Evaluate Safety and Pharmacokinetics of HLX70 in Healthy Adult Volunteers
Brief Title: Evaluate Safety and Pharmacokinetics of HLX70 in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategy.
Sponsor: Shanghai Henlius Biotech (Industry)
Collaborators: Hengenix Biotech Inc (Industry); Sanyou Biopharmaceuticals(Shanghai)Co., Ltd (Unknown); Shanghai ZJ Bio-Tech Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HLX70-001US; 255086 (Other: CRO study number)
Record Dates: First submitted 2022-04-29; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, Placebo-Controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HLX70 3 mg/kg or Placebo (Experimental): Random allocation to HLX70 3 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the HLX70.
  Interventions: Drug: HLX70; Drug: Placebo
- HLX70 10 mg/kg or Placebo (Experimental): Random allocation to HLX70 10 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the HLX70.
  Interventions: Drug: HLX70; Drug: Placebo
- HLX70 30 mg/kg or Placebo (Experimental): Random allocation to HLX70 30 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the HLX70.
  Interventions: Drug: HLX70; Drug: Placebo

INTERVENTIONS:
Drug: HLX70 — Single-dose, intravenous infusion
  Other Names: Recombinant Humanized Anti-S Protein Monoclonal Antibody for Injection
Drug: Placebo — Single-dose, intravenous infusion

SUMMARY:
A single-center, randomized, double-blind, placebo-controlled, dose escalation, phase I clinical study to evaluate safety and pharmacokinetics of HLX70 in healthy adult volunteers

DETAILED DESCRIPTION:
A randomized, double-blind, single-dose by intravenous administration, placebo-controlled, dose escalation, first-in-human study is proposed to evaluate the safety, PK, and immunogenicity of HLX70 in healthy subjects. We plan to enroll 8 subjects in each of the 3 dose cohorts at 3 mg/kg, 10 mg/kg, and 30 mg/kg, of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the investigational product (IP). A total of 24 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with voluntary signing of the informed consent form (ICF);
2. Healthy males or females aged ≥ 18 and ≤ 60 years at the time of signing the ICF;
3. Subjects with body weight ≥ 50 kg and body mass index (BMI) must be higher than 18.5 kg/m2 and lower than 30 kg/m2 at screening visit ;
4. Subjects who are determined to be in good health according to medical history, normal (site normal ranges to be followed) or abnormal but clinically insignificant physical examination, vital signs, ECG, laboratory test results (including hematology, serum chemistry, coagulation function, urinalysis, etc.), and investigator's clinical judgment (CTCAE grade 1 of triglycerides and uric acid is permitted). One re-test allowed per investigator discretion to confim result.
5. Subject who agrees that he and his spouse or partner will use reliable contraception for 9 months after administration.

Exclusion Criteria:

1. Subjects with the lab-confirmed medical history of COVID-19, including nucleic acid (PCR testing of nasopharyngeal samples) tested positive or antibody IgG/IgM tested positive.
2. Subjects with the novel onset of pyrexia/cough/shortness of breath/diarrhea or history of contact with confirmed COVID-19 individuals (positive for SARS-CoV-2 nucleic acid) within the 14 days before randomization.
3. Subjects who are known to have chronic obstructive pulmonary disease (COPD), cirrhosis of liver, cardiac failure or any condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being.
4. Subjects with pneumonia or tuberculosis (TB) suggested by chest X-Ray.
5. Subjects with previous exposure to a mAb or any other biological agents in 6 months before screening.
6. Subjects with previous exposure to vaccines in 3 months before screening, or who plans to receive vaccination during the study period or in 3 months after the study.
7. Subjects with previous participation in clinical trials receiving investigational drug/comparator within the longer of 30 days or 5 half-lives before screening.
8. Subjects who are known to have a history of allergy to any mAb, biological product, protein product, or the ingredient of the IP.
9. Subjects with positive test result(s) for hepatitis B virus (positive for HBsAg or positive for HBcAb and HBV-DNA), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, or treponema pallidum.
10. Subjects who are known to have a history of psychotropic drug abuse, alcoholism, or drug addiction within the last year.
11. Subjects with a history of a blood donation within 3 months before screening.
12. Subjects with the use of any prescription drug, OTC drug, or traditional Chinese medicine in 14 days before screening.
13. Females who are pregnant or breastfeeding
14. Other factors that the Investigator deems inappropriate for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-09 (Estimated); Primary Completion 2021-09-06 (Estimated); Study Completion 2021-09-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events, serious adverse event and infusion-related reactions as assessed by CTCAE v5.0 | up to 92 days.
  Safety follow-up: All subjects in the study will undergo safety follow-up within 92 days after administration and receive routine laboratory tests on day 2, day 3, day 8, day 15, day 22 and day 29 post administration (see the study procedures for details). A telephone follow-up will be followed every week until day 92 (day 1 is defined as the day of IP infusion). For a subject suffering AE during the observation period, follow-up shall be continued until the AE returns to the baseline or it is stable from getting worse.
Safety evaluation- proportion of subjects undergoing DLT events | Days 1 to 7.
  The proportion of subjects undergoing DLT events

SECONDARY OUTCOMES:
PK parameters-Areas under the concentration-time curves | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Maximum measured concentration | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Time from dosing to maximum measured concentration | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Terminal phase elimination rate constant | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Terminal phase elimination half life | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Clearance | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Volume of distribution during terminal phase and at steady state | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
PK parameters-Mean residence time | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
  PK blood sampling points: All subjects in the study will participate in the PK study. PK blood sampling timepoints: pre-infusion, immediately post-infusion, and 3 h, 6 h, 10 h, 24 h(Day 2), 48 h (day 3) , 96 h (day 5), 168 h (day 8) , 240h (day 11) , 336 h (day 15), 504 h (day 22) , 672 (day 29) , 1008 h (day 43) ,1344 h (day 57), 1680 h (day 71) , and 2184 h (day 92), after HLX70 infusion. There are a total of 17 blood sampling time points.
Anti-drug antibody | pre-infusion and Days 15, 29, 57 and 92.
  Blood sampling time points for immunogenicity: Blood samples for anti-drug antibody (ADA) testing will be collected at pre-infusion and on day 15, day 29, day 57, and day 92 after administration; positive ADA samples will be tested for neutralizing antibody (NAb).

IPD SHARING:
Plan to Share IPD: No